CLINICAL TRIAL: NCT00258427
Title: Hematopoietic Stem Cell Transplantation in High Risk Patients With Fanconi Anemia MT2002-02
Brief Title: Hematopoietic Stem Cell Transplantation in High Risk Patients With Fanconi Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002LS014; MT2002-02 (Other: Blood and Marrow Transplantation Program); 0202M18741 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Antilymphocyte Serum; Filgrastim; Granulocyte Colony-Stimulating Factor; Busulfan; Cyclophosphamide; fludarabine phosphate; Methylprednisolone; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Marrow Isolex (Experimental): Bone marrow processed using Isolex300i
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Biological: Hematopoietic stem cell transplantation
- USB arm (Experimental): No processing
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Biological: Hematopoietic stem cell transplantation
- Marrow Clinimacs (Experimental): Bone marrow processed using CliniMACS system
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Biological: Hematopoietic stem cell transplantation
- Sibling without CliniMacs (Experimental): Sibling donor without the use of CliniMACS system
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — Given 15 mg/kg/day intravenously every 12 hours on Days -5 through -1.
  Other Names: ATG
Biological: filgrastim — given 5 mcg/kg/day intravenously on Day 1 (continue until absolute neutrophil count (ANC) ≥2.5 x 10^9/L)
  Other Names: G-CSF
Drug: busulfan — Busulfan 0.8 mg/kg intravenously (IV) every 12 hours on Days -7 and -6 (1.0 mg/kg IV if <4 years old)
  Other Names: Busulfex
Drug: cyclophosphamide — 10 mg/kg intravenously (IV) on Days -5 through -2.
  Other Names: Cytoxan
Drug: fludarabine phosphate — 35 mg/m^2 intravenously (IV) on Days -5 through -2.
  Other Names: Fludara
Drug: methylprednisolone — 1 mg/kg intravenously (IV) every 12 hours on Days -5 through -1.
  Other Names: Medrol
Biological: Hematopoietic stem cell transplantation — Infused on Day 0 - Donor bone marrow or umbilical cord blood will be collected in the usual sterile manner using established parameters determined by the National Marrow Donor Program.
  Other Names: HSCT

SUMMARY:
RATIONALE: A bone marrow or umbilical cord blood transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Giving combination chemotherapy before a donor stem cell transplant may make the transplant more likely to work. This may be an effective treatment for patients with high risk Fanconi's anemia.

PURPOSE: This clinical trial is studying how well combination chemotherapy works in treating high risk patients who are undergoing a donor stem cell transplant for Fanconi's anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the incidence of neutrophil engraftment is acceptable in high-risk patients with Fanconi's anemia treated with busulfan, cyclophosphamide, fludarabine, and antithymocyte globulin followed by allogeneic hematopoietic stem cell transplantation.

Secondary

* Determine the tolerability of mycophenolate mofetil in these patients.
* Determine the incidence of acute and chronic graft-vs-host disease in patients treated with this regimen.
* Determine the incidence of major infections in patients with a history of major infections treated with this regimen.
* Determine the incidence of relapse in patients with refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, or acute myeloid leukemia treated with this regimen
* Determine the probability of 1-year survival of patients treated with this regimen.

OUTLINE: Patients are stratified according to donor/recipient HLA type (identical vs other).

* Cytoreductive combination chemotherapy: Patients receive busulfan intravenously (IV) over 2 hours twice daily on days -7 and -6 and cyclophosphamide IV over 2 hours and fludarabine IV over 30 minutes once daily on days -5 to -2.
* Graft failure prophylaxis: Patients receive methylprednisolone IV twice daily on days -5 to 30 and anti-thymocyte globulin IV over 4-6 hours twice daily on days -5 to -1.
* Graft-vs-host disease prophylaxis: Patients receive cyclosporine IV over 2 hours twice daily on days -3 to 100 (if patient has a matched sibling donor) or days -3 to 180 (if patient has another donor type). Patients also receive mycophenolate mofetil orally or IV twice daily on days -3 to 45.
* Allogeneic hematopoietic stem cell transplantation (HSCT): Patients undergo allogeneic HSCT (using bone marrow or umbilical cord blood) on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be <45 years of age with a diagnosis of Fanconi anemia with:

  * Biallelic BRCA2 mutations, or
  * Aplastic anemia, or advanced myelodysplastic syndrome (MDS) (MDS with ≥5% blasts), or acute leukemia who are ineligible for total body irradiation. Aplastic anemia is defined as having at least one of the following (with or without cytogenetic abnormalities): platelet count <20 * 10^9, - absolute neutrophil count (ANC) <5 * 10^8/L, - Hgb <8 g/dL
* Patients must have an HLA-A, B, DRB1 identical or 1 antigen mismatched related or unrelated BM donor or have an HLA-A, B, DRB1 identical, 1 antigen or 2 antigen mismatched related or unrelated umbilical cord blood (UCB) donor. Patients and donors will be typed for HLA-A and B using serological level typing and for DRB1 using high resolution molecular typing.
* Adequate major organ function including:

  * Cardiac: ejection fraction >45%
  * Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites, no cirrhosis)
  * Karnofsky performance status >70% or Lansky >50%
* Women of child bearing potential must be using adequate birth control and have a negative pregnancy test.

Exclusion Criteria:

* Active CNS leukemia at time of HSCT.
* Active uncontrolled infection within one week of hematopoietic stem cell transplant (HSCT).
* Pregnant or lactating female.

Donor Inclusion Criteria:

* Donor must be in good health based on review of systems and results of physical examination.
* Donor must have a normal hemoglobin, white count, platelet count and partial thromboplastin time (PTT), and a negative diepoxybutane (DEB) test.
* HIV-NAT negative, HTLV-1, HTLV-2 negative, Hepatitis B and C negative.
* Female donors of childbearing potential must have a negative pregnancy test.
* Unrelated donors must agree to peripheral blood stem cell (PBSC) donation

Donor Exclusion Criteria:

* Donor is a lactating female.

Max Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2002-03-26 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Marrow Clinimacs: Bone marrow processed using CliniMACS
- Sibling withoutCliniMACS: sibling donor without use of CliniMACS system
Period: Overall Study
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Started | 3 | 8 | 2 | 1
Completed | 3 | 8 | 2 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS | Total
Number analyzed (Participants) | 3 | 8 | 2 | 1 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 8 | 2 | 1 | 12
  Between 18 and 65 years | 2 | 0 | 0 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 5
  Male | 2 | 5 | 1 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 2 | 1 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 3
  White | 3 | 2 | 2 | 1 | 8
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 8 | 2 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Graft Failure
Description: Graft failure is defined as absolute neutrophil count( ANC ) <5 x 10^8/L by day 30.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 1 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Experiencing Chronic Graft-Versus-Host Disease
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cellsinto a foreign host.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Chronic Graft-Versus-Host Disease
Description: as for outcome 2
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Acute Graft-Versus-Host Disease
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Acute Graft-Versus-Host Disease
Description: as for outcome 4
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Relapse
Description: Patients with leukemia will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 0 | 2 | 1 | 0

7. Secondary Outcome: Number of Participants Experiencing Overall Survival
Description: Overall Survival - Number of patients alive at 1 year post transplant
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 1 | 4 | 1 | 1

8. Secondary Outcome: Number of Participants Experiencing Major Infections
Description: Number of participants experiencing Major Infections by the end of treatment
Time Frame: Day 1 through 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
Number analyzed (Participants) | 3 | 8 | 2 | 1
Participants | 3 | 8 | 2 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Marrow Isolex | USB Arm | Marrow Clinimacs | Sibling withoutCliniMACS
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/8 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/8 | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 7/8 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marrow Isolex (N=3) | USB Arm (N=8) | Marrow Clinimacs (N=2) | Sibling withoutCliniMACS (N=1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Primary Graft Failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marrow Isolex (N=3) | USB Arm (N=8) | Marrow Clinimacs (N=2) | Sibling withoutCliniMACS (N=1)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Tube Placement (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest Xray (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dialysis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Rash with Eosinophilia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Engraftment syndrome (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Eosinophilic gut (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (18) | 6 (18) | 1 (1) | 1 (1)
Intubation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pleuracentesis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (10) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Primary Graft Failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unresponsive (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Veno occlusive disease (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT00258427/Prot_SAP_000.pdf